CLINICAL TRIAL: NCT00909155
Title: Non-Invasive Brain Imaging Techniques That Predict Antidepressant Responsiveness and Provide Insights Into the Mechanism of Action of Venlafaxine ER vs. Fluoxetine
Brief Title: Brain Imaging Techniques That Predict Antidepressant Responsiveness
Acronym: WyethKolden
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 0600B-100953; 2001-294 (Other: HS IRB)
Record Dates: First submitted 2009-05-18; First posted 2009-05-27 (Estimated); Results first posted 2014-12-15 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-07

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Venlafaxine Hydrochloride; Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Depressed; Venlafaxine treatment (Active Comparator): Currently depressed subjects; Randomized medication treatment with Venlafaxine extended release tablets (Venlafaxine ERT). Dosage 75-300mg/day for up to 6 months.
  Interventions: Drug: Venlafaxine ERT
- Depressed; Fluoxetine treatment (Active Comparator): Currently depressed subjects; Randomized medication treatment with Fluoxetine tablets. Dosage 20-80mg/day for up to 6 months.
  Interventions: Drug: Fluoxetine
- Control (No Intervention): Non-psychiatric subjects with no past or current history of depression. Subjects will receive no medication

INTERVENTIONS:
Drug: Venlafaxine ERT — Titrated to a minimum dose of 75mg. Further titration based on clinician assessment at followup visits. Intervention to continue through completion of study (180 days). Initial titration: Days 1-7: 37.5 mg; Days 7-14: 75 mg; Days 15-180: 75-300mg based on clinician assessment. Titration rate is a maximum of 75mg/7d.
  Other Names: Effexor ER
  Arms: Depressed; Venlafaxine treatment
Drug: Fluoxetine — Titrated to a minimum dose of 20mg. Further titration based on clinician assessment at followup visits. Intervention to continue through completion of study (180 days). Initial titration: Days 1-7: 20mg; Days 7-14: 20mg; Days 15-180: 20-80mg based on clinician assessment. Titration rate is a maximum of 20mg/7d
  Other Names: Prozac
  Arms: Depressed; Fluoxetine treatment

SUMMARY:
Do functional brain changes occur during Venlafaxine ER (extended release) versus Fluoxetine treatment and do changes in selective structures, such as the amygdala, predict treatment response?

DETAILED DESCRIPTION:
This is a single site, controlled, double-blind study of outpatients. There are two arms:

1. Forty participants who have a current Diagnostic and Statistical Manual of Mental Disorders, 4th edition, text revised (DSM-IV-TR) diagnosis of Major Depression will be recruited. These subjects will be randomized to receive one of two antidepressant medications: Fluoxetine or Venlafaxine ER for the duration of the study. Subjects will gradually be titrated onto the medications and will be seen in the clinic up to 18 times for medication checks, to monitor side effects and depressive symptoms, including suicidal ideation. In the event of suicidal ideation, subjects will be withdrawn from the study and referred for immediate treatment.
2. Twenty normal control subjects with no current or past DSM-IV-TR diagnosis and will receive no medication. Normal control subjects will have up to 5 visits while in the study.

Subjects will contact study staff to complete a phone screen and then eligible subjects will complete a clinic screen. Subjects will then be scheduled to attend the magnetic resonance imaging (MRI) simulation visit and if subjects continue to meet entrance criteria, they will be scheduled for the first MRI. Following the first MRI, subjects in the medication conditions will begin receiving medication.

All subjects will undergo 3 functional magnetic resonance imaging (fMRI)s during the study: at the beginning of the study, approximately 8 weeks and 26 weeks later. During the MRI, subjects will view slides with positive and negative emotional content. Subjects will complete various clinical interviews or rating scales assessing mood and side effects at each of the visits.

ELIGIBILITY:
Inclusion Criteria:

* Intervention Group:

  * Right-handed,
  * Be able to lie still on their back for about 120 minutes,
  * Meet DSM-IV criteria for major depression (single or recurrent),
  * Have had depressive symptoms for at least 1 month prior to screen visit,
  * Must score an 18 or above on the Hamilton-D at both the initial screening visit and first fMRI scanning session,
  * Able to understand and speak English.
* Control Group: same as above with the exception of no diagnosis of psychiatric disorder.

Exclusion Criteria:

* Any history of seizures,
* Current medical disorders that might make interpretation of scan data difficult,
* Diabetes requiring insulin treatment,
* A serious heart disorder or subjects who have had a heart attack within the last 3 months,
* Subjects who meet DSM-IV criteria for alcohol/drug abuse or dependence within the last six months,
* Other current DSM-IV Axis I or Axis II diagnoses,
* A personal or family history of bipolar disorder,
* Current use of medication that affects central nervous system (CNS) function,
* Participation in the last 30 days in a clinical study involving an investigational drug,
* A subject with metallic implants, such as prostheses, shrapnel or aneurysm clip-S, or persons with electronic implants, such as cardiac pacemakers. The magnetic field generated by the MRI machine can cause a displacement or malfunctioning of these devices.
* A subject who is claustrophobic,
* Female subjects who are pregnant,
* A subject at serious risk for suicide,
* Diagnosis of cancer in the past 3 years and/or has active neoplastic disease,
* Nonresponse to 2 adequate trials of antidepressant treatment,
* Nonresponse to 2 adequate trials of an empirically supported psychotherapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2002-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Kolden, Ph.D., Principal Investigator — University of Wisconsin Madison Psychiatry Department; Michael Peterson, MD, Ph.D., Principal Investigator — University of Wisconsin Madison Psychiatry Department
Locations (1):
- University of Wisconsin Madison Psychiatry Department, Madison, Wisconsin, United States

REFERENCES:
- [Result] Heller AS, Johnstone T, Peterson MJ, Kolden GG, Kalin NH, Davidson RJ. Increased prefrontal cortex activity during negative emotion regulation as a predictor of depression symptom severity trajectory over 6 months. JAMA Psychiatry. 2013 Nov;70(11):1181-9. doi: 10.1001/jamapsychiatry.2013.2430. PMID 24173657
- [Result] Heller AS, Johnstone T, Light SN, Peterson MJ, Kolden GG, Kalin NH, Davidson RJ. Relationships between changes in sustained fronto-striatal connectivity and positive affect in major depression resulting from antidepressant treatment. Am J Psychiatry. 2013 Feb;170(2):197-206. doi: 10.1176/appi.ajp.2012.12010014. PMID 23223803
- [Result] Light SN, Heller AS, Johnstone T, Kolden GG, Peterson MJ, Kalin NH, Davidson RJ. Reduced right ventrolateral prefrontal cortex activity while inhibiting positive affect is associated with improvement in hedonic capacity after 8 weeks of antidepressant treatment in major depressive disorder. Biol Psychiatry. 2011 Nov 15;70(10):962-8. doi: 10.1016/j.biopsych.2011.06.031. Epub 2011 Aug 25. PMID 21867991
- [Result] Heller AS, Johnstone T, Shackman AJ, Light SN, Peterson MJ, Kolden GG, Kalin NH, Davidson RJ. Reduced capacity to sustain positive emotion in major depression reflects diminished maintenance of fronto-striatal brain activation. Proc Natl Acad Sci U S A. 2009 Dec 29;106(52):22445-50. doi: 10.1073/pnas.0910651106. Epub 2009 Dec 22. PMID 20080793

RESULTS

PARTICIPANT FLOW:
Groups:
- Currently Depressed Subjects: Venlafaxine: Currently depressed subjects; Randomized medication treatment with Venlafaxine extended release tablets (Venlafaxine ERT).
  Venlafaxine ERT: Titrated to a minimum dose of 75mg. Further titration based on clinician assessment at followup visits. Intervention to continue through completion of study (180 days). Initial titration: Days 1-7: 37.5 mg; Days 7-14: 75 mg; Days 15-180: 75-300mg based on clinician assessment. Titration rate is a maximum of 75mg/7d.
- Currently Depressed Subjects: Fluoxetine: Currently depressed subjects; Randomized medication treatment with Fluoxetine
  Fluoxetine: Titrated to a minimum dose of 20mg. Further titration based on clinician assessment at followup visits. Intervention to continue through completion of study (180 days). Initial titration: Days 1-7: 20mg; Days 7-14: 20mg; Days 15-180: 20-80mg based on clinician assessment. Titration rate is a maximum of 20mg/7d
- Control (Non-psychiatric Subjects): Non-psychiatric subjects with no past or current history of depression. Subjects will receive no medication
Period: Overall Study
Arm/Group | Currently Depressed Subjects: Venlafaxine | Currently Depressed Subjects: Fluoxetine | Control (Non-psychiatric Subjects)
Started | 15 | 14 | 21
Completed | 12 | 9 | 14
Not Completed | 3 | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Currently Depressed Subjects: Venlafaxine: Currently depressed subjects; Randomized medication treatment with Venlafaxine ERT
  Venlafaxine ERT: Titrated to a minimum dose of 75mg. Further titration based on clinician assessment at followup visits. Intervention to continue through completion of study (180 days). Initial titration: Days 1-7: 37.5 mg; Days 7-14: 75 mg; Days 15-180: 75-300mg based on clinician assessment. Titration rate is a maximum of 75mg/7d.
- Total: Total of all reporting groups
Arm/Group | Currently Depressed Subjects: Venlafaxine | Currently Depressed Subjects: Fluoxetine | Control (Non-psychiatric Subjects) | Total
Number analyzed (Participants) | 15 | 14 | 21 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 14 | 21 | 50
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Data from the fluoxetine and venlafaxine groups were combined for analysis as individual groups not large enough to provide sufficient statistical power to identify treatment differences between groups.
  years | 30.74 (11.46) | 33.14 (10.71) | 31.31 (14.22) | 31.65 (12.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 13 | 29
  Male | 7 | 6 | 8 | 21
Region of Enrollment [Number; unit: participants]
  United States | 15 | 14 | 21 | 50

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression (HAM-D) and Anxiety (HAM-A) Rating Scales
Description: Hamilton Depression rating scale is a clinician assessment tool to measure severity of depression symptoms. Minimum score is 0 (no symptoms); maximum score is 52 (severe symptoms of depression).
  Hamilton Anxiety rating scale is a clinician assessment tool to measure severity of anxiety symptoms. Minimum score is 0 (no symptoms); maximum score is 56 (severe symptoms of anxiety).
Time Frame: Study entry, 2 months, and at end of study (6 mos)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Currently Depressed Subjects: Venlafaxine | Currently Depressed Subjects: Fluoxetine | Control (Non-psychiatric Subjects)
Number analyzed (Participants) | 15 | 14 | 21
units on a scale
  HAMD T0 | 20.07 (1.94) | 21.36 (2.71) | 1 (1.55)
  HAMA T0 | 14.07 (3.37) | 15.57 (3.82) | NA (NA) — HAMA not collected on control subjects.
  HAMD 2months | 8.86 (4.5) | 10.15 (4.52) | 1.25 (1.34)
  HAMA 2months | 7.5 (4.55) | 8.54 (4.86) | NA (NA) — HAMA not collected on control subjects.
  HAMD 6months | 5 (3.67) | 7.33 (4.92) | 1.64 (1.22)
  HAMA 6months | 4.25 (3.36) | 5.89 (3.86) | NA (NA) — HAMA not collected on control subjects.

2. Primary Outcome: Functional Magnetic Resonance Imaging (fMRI) Response to an Emotional Regulation Task.
Description: Depressed participants were scanned while viewing a sequence of positive and negative images; they were instructed to enhance or supress their emotional response to the image or to continue to attend. To examine brain function when regulating negative affect, we created contrast maps for each participant at all 3 time points by subtracting the attend condition from the suppress condition in response to negative stimuli. Data from all 3 scan sessions were used to assess treatment-induced change in brain activity when regulating emotion. Analyses examining change using difference scores (end vs. starting points), we subtracted initial HAMD score from final HAMD score. For fMRI analyses, in a voxelwise manner, we subtracted initial negative suppress vs attend from final negative suppress vs attend.
  Control subjects were not depressed, repeat scans to assess change were not completed.
  Reported results are from BA10, one of our areas of interest.
Time Frame: At study entry, 2 months and end of study (6 months)
Population: Depressed subjects were treated with an SSRI or an SNRI, and assessed at 3 time points on an fMRI emotional response task. Differences in depression scores and changes in the fMRI responses were analyzed for changes to better understand the association between emotion regulation, depression, and treatment response.
Measure: Mean (Standard Deviation); unit: fMRI signal change
Groups:
- Depressed; Venlafaxine Treatment: Currently depressed subjects; Randomized medication treatment with Venlafaxine extended release tablets (Venlafaxine ERT). Dosage 75-300mg/day for up to 6 months.
  Venlafaxine ERT: Titrated to a minimum dose of 75mg. Further titration based on clinician assessment at followup visits. Intervention to continue through completion of study (180 days). Initial titration: Days 1-7: 37.5 mg; Days 7-14: 75 mg; Days 15-180: 75-300mg based on clinician assessment. Titration rate is a maximum of 75mg/7d.
  12 subjects completed the treatment, and both the 2month and 6month fMRI scans.
- Depressed; Fluoxetine Treatment: Currently depressed subjects; Randomized medication treatment with Fluoxetine tablets. Dosage 20-80mg/day for up to 6 months.
  Fluoxetine: Titrated to a minimum dose of 20mg. Further titration based on clinician assessment at followup visits. Intervention to continue through completion of study (180 days). Initial titration: Days 1-7: 20mg; Days 7-14: 20mg; Days 15-180: 20-80mg based on clinician assessment. Titration rate is a maximum of 20mg/7d.
  9 subjects completed the treatment, and both the 2month and 6month fMRI scans.
- Control: Non-psychiatric subjects with no past or current history of depression. Subjects will receive no medication.
  Control subjects did not complete the 2month and 6month fMRI scans since no depression was present, no treatment given, and no change in mood state expected.
  As such, no change in depression score could be calculated to provide a comparable measure in this group analysis. This analysis looked for functional imaging findings that correlated with improvement in depression symptoms.
Arm/Group | Depressed; Venlafaxine Treatment | Depressed; Fluoxetine Treatment | Control
Number analyzed (Participants) | 12 | 9 | 0
fMRI signal change | -0.042666667 (0.291892646) | 0.0414 (0.332904397) |

ADVERSE EVENTS:
Groups:
- Currently Depressed Subjects; Venlafaxine: Currently depressed subjects; Randomized medication treatment with Venlafaxine ERT.
  Venlafaxine ERT: Titrated to a minimum dose of 75mg. Further titration based on clinician assessment at followup visits. Intervention to continue through completion of study (180 days). Initial titration: Days 1-7: 37.5 mg; Days 7-14: 75 mg; Days 15-180: 75-300mg based on clinician assessment. Titration rate is a maximum of 75mg/7d.
- Currently Depressed Subjects; Fluoxetine: Currently depressed subjects; Randomized medication treatment with Fluoxetine
  Fluoxetine: Titrated to a minimum dose of 20mg. Further titration based on clinician assessment at followup visits. Intervention to continue through completion of study (180 days). Initial titration: Days 1-7: 20mg; Days 7-14: 20mg; Days 15-180: 20-80mg based on clinician assessment. Titration rate is a maximum of 20mg/7d
Arm/Group | Currently Depressed Subjects; Venlafaxine | Currently Depressed Subjects; Fluoxetine | Control (Non-psychiatric Subjects)
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14 | 0/21
Other Adverse Events (participants affected / at risk) | 0/15 | 0/14 | 0/21

LIMITATIONS AND CAVEATS:
Relatively small number of subjects. Not powered statistically to determine if either treatment arm (fluoxetine or venlafaxine) is superior.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No